CLINICAL TRIAL: NCT07124169
Title: Therapeutic Effects of Kinesiotape in the Management of Gonarthrosis: A Randomized Controlled Approach
Brief Title: Therapeutic Effects of Kinesiotape in the Management of Gonarthrosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenerbahce University (Other)
Responsible Party: Principal Investigator, Burcu AKKURT, assistant professor, Fenerbahce University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2015-17/04
Record Dates: First submitted 2025-08-05; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Gonarthrosis
Keywords: gonarthrosis; kinesiotape; home exercises
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Athletic Tape

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Kinesiotape+home exercise) (Experimental): The taping procedure was repeated once a week, starting from the first week, for a total of 6 sessions. Mechanical correction technique and Ligament/Tendon correction technique, as kinesiotape application, were performed. ). A 6-week home exercise program was given to both the taping and control groups, three sessions per week. An individualized home exercise program was planned, considering EULAR and ACR recommendations. Each participant was given a structured home exercise program for approximately 30 minutes per day, at least 3 days a week. The program included moderate-intensity aerobic exercises (e.g., walking) and muscle-strengthening exercises targeting the quadriceps and hamstring muscles, along with flexibility and balance exercises. ).
  Interventions: Other: Kinesiotape + home exercise
- control (home exercise ) (Active Comparator): A 6-week home exercise program was given to both the taping and control groups, three sessions per week. An individualized home exercise program was planned, considering EULAR and ACR recommendations. Each participant was given a structured home exercise program for approximately 30 minutes per day, at least 3 days a week. The program included moderate-intensity aerobic exercises (e.g., walking) and muscle-strengthening exercises targeting the quadriceps and hamstring muscles, along with flexibility and balance exercises.
  Interventions: Other: Home exercise

INTERVENTIONS:
Other: Kinesiotape + home exercise — Kinesiotaping will be applied to the knee once weekly for 6 weeks. In addition, participants will perform a structured home exercise program three times per week, including strengthening, stretching, and balance exercises.
  Arms: Experimental (Kinesiotape+home exercise)
Other: Home exercise — In addition, participants will perform a structured home exercise program three times per week, including strengthening, stretching, and balance exercises.
  Arms: control (home exercise )

SUMMARY:
This randomized controlled trial evaluated the effectiveness of kinesiotaping in addition to exercise for patients with knee osteoarthritis (gonarthrosis). Thirty-eight participants aged 45 to 65 were randomly assigned to two groups: one group performed a structured home exercise program three times weekly for 6 weeks, while the other group performed the same program and also received kinesiotaping once weekly. Outcomes included pain, stiffness, balance, and quality of life. Both groups demonstrated significant improvement; however, the kinesiotaping plus exercise group showed greater gains in pain reduction, mobility, and daily activities. These findings suggest that kinesiotaping combined with exercise may provide superior benefits compared with exercise alone in individuals with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* having a diagnosis of primary gonarthrosis according to ACR classification criteria,
* being between 45 and 65 years of age,
* having a radiological diagnosis of gonarthrosis between Kellgren-Lawrence stage 1-3 ,
* signing the informed consent

Exclusion Criteria:

* presence of a neurological disorder affecting muscle strength or balance,
* history of any surgical operation on the knee, hip or spine,
* physiotherapy or injections for the knee within the previous year,
* presence of systemic conditions such as diabetes mellitus, vertigo, visual problems,
* history of severe trauma within the previous year

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2015-11 (Actual); Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | From enrollment to the end of treatment at 6 weeks
  WOMAC consists of 24 questions in total (pain 5, joint stiffness 2, functional status 17). Each question was scored on a scale of 1-5. A high score indicates poor health, while a low score indicates good health.

SECONDARY OUTCOMES:
Visual Analogue Scale (VAS) | From enrollment to the end of treatment at 6 weeks
  VAS, which ranges from 0 to 10, is used to assess pain levels. A score of 0 represents no pain, while 10 indicates the most severe, unbearable pain. Participants were instructed to indicate their perceived pain level by marking a 10 cm straight line, and the corresponding value was recorded in centimeters.
Berg Balance Scale (BBS) | From enrollment to he end of treatment at 6 weeks.
  BBS is a test consisting of 14 items used to evaluate the functional balance of individuals. The application time is approximately 15-20 minutes, and the following materials are needed: a ruler, a stopwatch, a chair, a step, and an area suitable for 360-degree rotation. Each item is evaluated on a scale of 0-4 points based on the individual's ability to perform the given task independently and correctly. The total score is 56. A score between 0-20 indicates severe balance impairment, between 21-40 indicates acceptable balance, and between 41-56 indicates good balance.
Short Form (SF-36) | From enrollment to the end of treatment at 6 weeks
  The SF-36 questionnaire was developed to assess quality of life. A total of 8 sub-parameters, including pain, social functioning, energy/vitality, emotional role difficulties, physical role difficulties, physical functioning, general health perception, and mental health, are examined

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to concerns regarding patient confidentiality and data privacy

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-11-25): https://cdn.clinicaltrials.gov/large-docs/69/NCT07124169/Prot_SAP_000.pdf